CLINICAL TRIAL: NCT02525549
Title: Comparative Safety and Bioequivalence of Two Treatments in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-817
Record Dates: First submitted 2015-08-14; First posted 2015-08-17 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test product (Experimental): Adapalene and Benzoyl Peroxide Gel
  Interventions: Drug: Adapalene and Benzoyl Peroxide Gel
- Reference product (Active Comparator): Adapalene and Benzoyl Peroxide Gel (Reference)
  Interventions: Drug: Adapalene and Benzoyl Peroxide Gel (Reference)
- Placebo product (Placebo Comparator): Placebo gel
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Adapalene and Benzoyl Peroxide Gel
  Arms: Test product
Drug: Adapalene and Benzoyl Peroxide Gel (Reference)
  Arms: Reference product
Drug: Placebo gel
  Arms: Placebo product

SUMMARY:
The purpose of this study is to compare the safety and bioequivalence of Perrigo's product to an FDA approved product for the treatment acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female subjects, 12 to 40 years of age (inclusive), with a clinical diagnosis of at least moderate facial acne vulgaris
* Inflammatory lesion (papules and pustules) count of 20 to 50 (inclusive)
* Non-inflammatory (open and closed comedones) lesion count of 25 to 100 (inclusive)
* No more than two nodulocystic lesions (i.e., nodules and cysts) on the face including those present on the nose, were enrolled.
* Subjects must also have had a Baseline IGA score of 3 or 4 on a severity scale of 0 to 4 to be enrolled.

Exclusion Criteria:

* Subjects who are pregnant, nursing, or planning a pregnancy within the study participation period.
* Presence of more than 2 facial Nodulocystic lesions (i.e. nodules and cysts)
* Subjects with active cystic acne or Polycystic Ovarian Syndrome
* Presence of any other facial skin condition that, in the Investigator's opinion, might interfere with acne vulgaris diagnosis and/or evaluations (e .g., on the face: rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acneform eruptions caused by medications, steroid acne, steroid folliculitis, or bacterial folliculiti s).
* Excessive facial hair (e.g. beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of acne vulgaris.
* Acne conglobata, acne fulminan s, or secondary acne (chloracne, drug-induced acne, etc.)
* Use of antipruritics including antihistamine, within 24 hours prior to all study visits (Visit l/Baseline through Visit 4).
* Use of medicated make-up throughout the study and significant change in the use of consumer products within 30 days of study entry and throughout the study (other than study supplied cleanser and lotion).
* Use within 6 months prior to baseline or during the study of oral retinoids (e.g. Accutane"') or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed).
* Use within 1 month prior to baseline or during the study of therapeutic vitamin D supplement (multivitamins are allowed).
* Use within 1 month prior to baseline or during the study of 1) systemic sterOids', 2) systemic antibiotics, 3) systemic treatment for acne vulgaris (other than oral retinoids which require a 6-month washout), or 4) systemic anti-inflammatory agents". (' Intranasal and inhaled corticosteroids do not require a washout and may be used throughout the study if at a stable and standard dose. "Subjects may use Acetaminophen for pain relief, as needed, throughout the study)
* Use within 14 days prior to baseline or during the study of 1) topical sterOids, 2) topical retinoids, 3) topical acne treatments including over-the-counter preparation (e.g. azelaic acid,etc.) 4)a-hydroxy/glycolic acid, 5) benzoyl peroxide, 6) topical anti-inflammatory agents, or 7) topical antibiotics.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 903 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Product | Reference Product | Placebo Product
Started | 365 | 360 | 178
Completed | 330 | 307 | 159
Not Completed | 35 | 53 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference Product | Placebo Product | Total
Number analyzed (Participants) | 365 | 360 | 178 | 903
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.9 (6.25) | 20.4 (6.96) | 19.5 (6.55) | 20.0 (6.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 213 | 103 | 515
  Male | 166 | 147 | 75 | 388
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 70 | 59 | 27 | 156
  Not Hispanic or Latino | 295 | 301 | 151 | 747
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 1 | 7
  Asian | 17 | 19 | 7 | 43
  Native Hawaiian or Other Pacific Islander | 4 | 2 | 1 | 7
  Black or African American | 73 | 87 | 34 | 194
  White | 259 | 245 | 132 | 636
  More than one race | 6 | 3 | 0 | 9
  Unknown or Not Reported | 4 | 0 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline to Day 84 in Inflammatory (Papules and Pustules) Lesions
Time Frame: 84 days
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: percent change of lesion counts
Arm/Group | Test Product | Reference Product | Placebo Product
Number analyzed (Participants) | 268 | 247 | 134
percent change of lesion counts | 61.07 (36.6) | 65.58 (28.42) | 41.63 (28.05)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority — provides 85% power of success; Fieller's method; Equivalence ratio = 93.12, 90% CI 2-sided [88.6 to 102.00]

2. Primary Outcome: Mean Percent Change From Baseline to Day 84 in Non-inflammatory (Open and Closed Comedones) Lesions
Time Frame: 84 days
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: percent change of lesion counts
Arm/Group | Test Product | Reference Product | Placebo Product
Number analyzed (Participants) | 268 | 247 | 134
percent change of lesion counts | 54.33 (32.00) | 55.06 (32.62) | 36.40 (38.61)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority — provides 85% power of success; Fieller's method; Equivalence ratio = 98.7, 90% CI 2-sided [92.3 to 109.4]

ADVERSE EVENTS:
Time Frame: 84 Days
Arm/Group | Test Product | Reference Product | Placebo Product
All-Cause Mortality (participants affected / at risk) | 0/365 | 0/360 | 0/178
Serious Adverse Events (participants affected / at risk) | 0/365 | 2/360 | 2/178
Other Adverse Events (participants affected / at risk) | 0/365 | 0/360 | 0/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=365) | Reference Product (N=360) | Placebo Product (N=178)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2012-10-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT02525549/Prot_001.pdf
  • Statistical Analysis Plan (2012-10-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT02525549/SAP_000.pdf